CLINICAL TRIAL: NCT02543957
Title: A Prospective Study of the Factors Associated With Increased Risk of Bacteremia and Cholangitis in ERCP With Cholangioscopy
Brief Title: Factors Associated With Increased Risk of Bacteremia and Cholangitis in ERCP With Cholangioscopy
Status: Withdrawn | Type: Observational
Why Stopped: Funding not received.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Othman, M.D. Director of Advanced Endoscopy Assistant Professor of Medicine - Gastroenterology Section, Baylor College of Medicine
Other Study IDs: H-37346
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Cholangitis; Bacteremia
Keywords: ERCP; Cholangitis; Bacteremia; Antibiotics
MeSH Terms: conditions — Cholangitis; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Cholangioscopy — All patients will receive pre-procedural antibiotics per protocol. A blood culture will be drawn from patients prior to the procedure (before antibiotics administration), 5 minutes after the procedure and 30 minutes after the procedure. Patients will be followed up for 7 days after the procedure for fever and or sepsis.

SUMMARY:
An Endoscopic retrograde cholangio pancreatography (ERCP) with cholangioscopy (endoscope to directly visualize the bile duct ) is a procedure (a small flexible tube that is inserted into the participants mouth to the participants stomach and into the participants liver to visualize the bile duct) that is usually performed in patients for the following purposes :

1. The removal of all stones from the participants bile duct (if present).
2. Acquiring a tissue sample biopsy from any common bile mass to examine (if present).
3. Acquiring tissue sample biopsy from common bile duct narrowing (if present). However this procedure is associated with an increase risk of infection compared with the standard ERCP (ERCP without cholangioscopy). Previous studies have shown that despite the administration of antibiotics prior to these procedures, infection still occurs. This leads to a suspicion that other factors may be the cause in these infections. Factors such as age, race, gender and ethnicity have not been fully explored yet. This study aims to examine these factors in addition to others in patients who are undergoing ERCP with cholangioscopy as part of their routine medical care. This examination will allow us to bring out if any of the above mentioned factors may be involved in the development of an infection after ERCP with cholangioscopy.

DETAILED DESCRIPTION:
ERCP with cholangioscopy is becoming a widespread technique to treat complicated choledocholithiasis, document CBD clearance after stone extraction and to assess biliary duct strictures. During the procedure, a large amount of water is used to irrigate the common bile duct in order to improve visualization. This can result in CBD distension and may increase the possibility of bacterial translocation and subsequent bacteremia or septicemia. According to the ASGE guidelines, antibiotic prophylaxis prior to ERCP is indicated when biliary duct obstruction is suspected prior to ERCP procedures . There are no current guidelines addressing antibiotics prophylaxis prior to ERCP with cholangioscopy. The investigators recent ACG funded prospective trial examining the risk of bacteremia in ERCP with cholangioscopy have shown the presence of bacteremia in 8.8% of patients undergoing ERCP with cholangioscopy, thus prompting the use of prophylactic antibiotics in patients undergoing these procedures. However the study was not powered to examine factors associated with increased bacteremia and infectious complications. In spite of the use of pre-procedural antibiotics in some of the published series, infectious complications such as cholangitis and sepsis were still reported after the procedure. In the landmark study by Chen et al, in which 297 patients prospectively underwent single-operator cholangioscopy in 15 referral centers across the US and Europe, nine patients developed cholangitis. Antibiotics administration prior to the procedures was left to the standard of practice at each participating institution and was not reported in this study. In a retrospective study by Kalaitzakis et al, nine out of 179 patients who underwent cholangioscopy for CBD stricture or treatment of CBD stones developed cholangitis. Cholangitis was fatal in one case and required prolonged hospitalization in the other case. All patients in this study had antibiotics prophylaxis prior to the procedure. Manta et al had one case of cholangitis in their series of 52 patients who underwent cholangioscopy for CBD stricture. Two patients out of 87 patients had cholangitis in the study by Osania et al., which prospectively included patients who underwent cholangioscopy for CBD stricture. The cholangitis rate in the previously mentioned studies ranged from 2% to 5%. This high rate of post procedure cholangitis in spite of the use of pre-procedural antibiotics suggest that post procedure antibiotics are of value in subsets of patients who will undergo ERCP with cholangioscopy. In the investigators preliminary data, bacteremia rate was significantly higher in patients with CBD strictures who had cholangioscopy with biopsies. It is possible that strictures could lead to colonization of biliary epithelium with bacteria. Obtaining biopsies may cause disruption of the endothelial barrier allowing bacterial translocation. In addition, cholangitis was seen in one patient in the investigators cohort who underwent laser lithotripsy for large stone. Choledocholithiasis is another source of bacterial colonization which could increase the risk of cholangitis after ERCP and cholangioscopy. The investigators protocol objective is to examine the factors that are potentially associated with increased frequency of bacteremia and subsequent infectious complication after ERCP with cholangioscopy in a setting of uniform pre-procedure antibiotics. The investigators hypothesize that biopsy of CBD strictures and Laser Lithotripsy are risk factors for increased rate of bacteremia and infectious complications after ERCP with cholangioscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18-80) who are undergoing ERCP with cholangioscopy to ensure the clearance of the CBD from stones.
2. Adult patients (18-80) who are undergoing ERCP with cholangioscopy for CBD stone removal using laser lithotripsy.
3. Adult patients (18-80) who are undergoing ERCP with cholangioscopy for CBD mass.
4. Adult patients (18-80) who are undergoing ERCP with cholangioscopy for tissue acquisition from CBD strictures with biopsies.

Exclusion Criteria:

1. Patients younger than 18 yrs old or older than 80 yrs.
2. Pregnant patients.
3. Patient with ascending cholangitis, pneumonia or urinary tract infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants ages 18-80 will be recruited from patients undergoing an ERCP at the Baylor St Luke Medical center in Houston or at University of Texas Health Science Center at San Antonio. Both practices are university based practice and serve as a tertiary referral center for all complicated EUS and ERCP procedures in eastern Texas. Choledocholithiasis and its complications requiring ERCP are prevalent and represent a large share of this ERCP practice.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Examine the Incidence of new onset infectious complications | 7 days
  1- To examine the incidence and risk factors of new onset infectious complications such as fever, sepsis or cholangitis within one week after ERCP with cholangioscopy.

SECONDARY OUTCOMES:
Examine the incidence of bacteremia in patients undergoing ERCP with cholangioscopy | 7 days
  Existing prospective data have shown bacteremia in 8.8% of patients undergoing ERCP with cholangioscopy, thus promoting the use of prophylactic antibiotics in patients undergoing these procedures. Three blood withdrawals from the patient undergoing ERCP with Cholangioscopy. One blood withdrawal will be taken before the procedure (Cholangioscopy), the second one will be taken 5 minutes after the procedure and the last blood withdrawal will be taken 30 minutes after the procedure with an overall 30 cc blood withdrawn from each patient. Aseptic techniques will be taken to minimize the contamination of the blood sample by the skin flora. Patients with positive blood culture for bacteremia will be monitored and only patients with fever and evidence of sepsis or cholangitis will be treated with antibiotics. The patient will receive a phone questionnaire about adverse affects that might have happened after the procedure 24 hours after the procedure and 1 week after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Othman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States